CLINICAL TRIAL: NCT07196982
Title: Risk Factors for Intertrochanteric Femoral Fractures With Concomitant Lateral Wall Involvement in Elderly Women
Acronym: Fracture
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-HG-2025-107
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Intertrochanteric Femoral Fracture
Keywords: Intertrochanteric Fractures; Femoral Lateral Wall Fractures; Bone Mineral Density
MeSH Terms: conditions — Hip Fractures | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated Intertrochanteric Fracture: Postmenopausal women with intertrochanteric femoral fractures without lateral wall involvement.
- Intertrochanteric Fracture with Lateral Wall Involvement: Postmenopausal women with intertrochanteric femoral fractures with concomitant lateral wall involvement.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational retrospective case-control study. No experimental intervention is administered. All participants received standard surgical management for intertrochanteric femoral fractures according to clinical practice, including proximal femoral nail antirotation (PFNA) with or without additional lateral wall plate fixation. The study only compares clinical and radiological data between patients with isolated intertrochanteric fractures and those with concomitant lateral wall involvement.
  Groups: Intertrochanteric Fracture with Lateral Wall Involvement

SUMMARY:
This study aims to better understand the factors that increase the risk of a special type of hip fracture in older women, known as intertrochanteric femoral fractures with lateral wall involvement. Hip fractures are very common in elderly patients, especially in women after menopause, and can seriously affect independence, mobility, and quality of life.

Between January 2023 and February 2024, postmenopausal women who were admitted with intertrochanteric femoral fractures were studied. Among them, some patients had fractures only in the main hip area, while others had additional involvement of the lateral wall, an important supportive structure of the hip. Researchers collected information such as age, body mass index (BMI), bone mineral density (BMD), and bone metabolism markers.

The study found that women with lower BMI and lower bone mineral density at the hip and lumbar spine were more likely to have lateral wall involvement in their fractures. Age and blood markers of bone metabolism did not show a strong link.

Understanding these risk factors can help doctors improve preoperative evaluation, choose better surgical strategies, and recommend preventive measures such as bone health management and fall prevention. This may ultimately reduce complications, improve recovery, and support better long-term outcomes for elderly women with hip fractures.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women diagnosed with intertrochanteric femoral fractures.

History of low-energy trauma (e.g., fall from standing height).

Treated surgically with proximal femoral nail antirotation (PFNA) device, with or without lateral wall plate fixation.

Availability of complete demographic and clinical data (age, height, weight, bone mineral density, and bone turnover markers).

Eligible for retrospective case-control analysis.

Exclusion Criteria:

High-energy trauma (e.g., motor vehicle accidents).

Severe systemic comorbidities such as hepatic or renal failure, bone tumors, or endocrine disorders (e.g., hyperparathyroidism).

Use of medications affecting bone metabolism within 6 months before surgery.

Diagnosis of diabetes mellitus.

History of chronic smoking or alcohol abuse.

Inability to provide accurate anthropometric data (height and weight).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of postmenopausal women admitted to the Department of Orthopedics at the Second Affiliated Hospital of Soochow University between January 2023 and February 2024 with a diagnosis of intertrochanteric femoral fracture. A total of 49 patients were included after applying eligibility criteria. Of these, 29 had isolated intertrochanteric fractures and 20 had intertrochanteric fractures with concomitant lateral wall involvement. All patients underwent surgical fixation with proximal femoral nail antirotation (PFNA), with or without additional lateral wall plate fixation, according to clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Association between Bone Mineral Density, BMI, and Lateral Wall Involvement in Intertrochanteric Femoral Fractures | From hospital admission to postoperative BMD assessment (within 3 months of injury)
  The primary outcome is to determine whether reduced bone mineral density (BMD) and lower body mass index (BMI) are independent risk factors for lateral wall involvement in elderly women with intertrochanteric femoral fractures. Measurements include lumbar spine and hip BMD assessed by dual-energy X-ray absorptiometry (DXA) and BMI calculated from height and weight. Logistic regression analysis is used to evaluate associations between these factors and the presence of lateral wall fractures.

CONTACTS AND LOCATIONS:
Locations (1):
- The medical record system and imaging system of the Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Shi G, Hu Z, Xie Z, Gu J, Lu Q, Ling Z. Risk factors for intertrochanteric femoral fractures with concomitant lateral wall involvement in elderly women. Front Surg. 2025 Dec 18;12:1730094. doi: 10.3389/fsurg.2025.1730094. eCollection 2025. PMID 41488883